CLINICAL TRIAL: NCT02785406
Title: Role of the Orexin Receptor System in Stress, Sleep and Cocaine Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Peter McManus Charitable Trust (Other)
Responsible Party: Principal Investigator, Scott Lane, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-16-0120
Record Dates: First submitted 2016-05-19; First posted 2016-05-27 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Cocaine Use Disorder; Anxiety
Keywords: cocaine; sleep; anxiety; craving; addiction; orexin; cue reactivity; suvorexant; Belsomra
MeSH Terms: conditions — Anxiety Disorders; Behavior, Addictive | interventions — suvorexant; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- suvorexant (Experimental): Subjects will receive suvorexant (10 mg week 1, 20 mg week 2), once daily at 10 PM.
  Interventions: Drug: suvorexant
- Placebo (Placebo Comparator): Subjects will receive placebo once daily at 10 PM.
  Interventions: Drug: Placebo (for suvorexant)

INTERVENTIONS:
Drug: suvorexant — Subjects will receive suvorexant capsules (10 mg week 1, 20 mg week 2), once daily at 10 PM.
  Other Names: Belsomra
  Arms: suvorexant
Drug: Placebo (for suvorexant) — Subjects will receive placebo capsules once daily at 10 PM.
  Other Names: corn starch
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of a medication called suvorexant in reducing anxiety, improving sleep, and reducing cocaine cravings or cocaine use.

DETAILED DESCRIPTION:
Preclinical research has established important functions for the orexin system in mediating arousal/sleep, stress, and cue-induced reinstatement of drug taking (e.g., relapse). The role of stress/anxiety and drug cue reactivity in human drug relapse is well established, but to date, the role of the orexin system in modulating these phenomena has not been examined in humans with substance use disorders (e.g., cocaine). The goal of the present first-in-human study will be to examine the effects of an orexin antagonist (suvorexant) on interactions among stress/anxiety, sleep, and drug-cue reactivity. The study will utilize a battery of highly sensitive, drug-specific, laboratory measures of drug cue reactivity (a relapse risk model), and well-established metrics of stress/anxiety and sleep. The hypothesis is that antagonism of the orexin system will attenuate the link between (1) stress/anxiety and drug cue reactivity, and (2) sleep and drug cue reactivity. These results will elucidate a unique biochemical mechanism for understanding relapse, and provide a potential medication target for relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

* meet current DSM-5 criteria for cocaine use disorder (CUD) of at least moderate severity (≥4 symptoms)

Exclusion Criteria:

* current DSM-IV diagnosis of any psychoactive substance dependence other than cocaine, marijuana, or nicotine
* have a DSM-IV axis I psychiatric disorder or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe
* significant current suicidal or homicidal ideation
* medical conditions contraindicating administration of suvorexant (e.g., severe pulmonary disease, severe cardiovascular disease or clinically abnormal EEG, severe liver or kidney disease, seizure disorder, or sleep disorder - particularly narcolepsy)
* taking medications known to have significant drug interactions with the study medication(s) (e.g., MAO inhibitors, anticonvulsants, haloperidol, phenothiazines, anesthetics, and all sedatives)
* currently or recently (last 3 months) treated for substance use [other than cocaine or nicotine] or another psychiatric condition
* conditions of probation or parole requiring reports of drug use to officers of the court; (8) impending incarceration
* pregnant or nursing for female patients
* inability to read, write, or speak English [required for lab tasks and psychometric scales]
* unwillingness to sign a written informed consent form
* subjects with alcohol use disorders or are drinking > 7 alcoholic drinks per week. All subjects who are excluded will be given referral information to other local treatment programs.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Lane, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suvorexant | Placebo
Started | 10 | 10
Completed First Week | 10 | 10
Completed Second Week | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (6.7) | 46.6 (6.75) | 45.65 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 7 | 9 | 16
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cue Reactivity as Assessed by the Attention Bias (AB) Task
Description: The attention bias (AB) task is a saccade-based eye-tracking measurement, developed by the PI to assess attentional bias to drug cues. AB measures utilizing eye movements have produced moderate to robust effects for a broad class abused substances, including cocaine. The score ranges from 0 to 1. Higher scores indicate a worse outcome.
Time Frame: day 0
Population: Data were not collected for 1 in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 0.524 (0.0846) | 0.519 (0.107)

2. Primary Outcome: Cue Reactivity as Assessed by the Attention Bias (AB) Task
Description: as for outcome 1
Time Frame: day 7
Population: Data were not collected for one in the suvorexant arm and one in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | 0.443 (0.0694) | 0.492 (0.149)

3. Primary Outcome: Cue Reactivity as Assessed by the Attention Bias (AB) Task
Description: as for outcome 1
Time Frame: day 14
Population: Data were not collected for one in the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 0.488 (0.19) | 0.508 (0.0832)

4. Primary Outcome: Total Sleep as Assessed by the Misfit Shine Device
Description: Sleep activity is monitored with a 3-axis accelerometer inside the watch device (Misfit Shine), using a general heuristic based on time and motion. The device is waterproof and worn on the wrist 24 hrs per day. Data are downloaded to smartphone via Bluetooth.
Time Frame: day 0
Population: Data were not collected for one in the suvorexant arm and 5 in the placebo arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 9 | 5
hours | 8.18 (2.17) | 8.05 (2.72)

5. Primary Outcome: Total Sleep as Assessed by the Misfit Shine Device
Description: as for outcome 4
Time Frame: day 2
Population: Data were not collected for 2 in the suvorexant arm and 4 in the placebo arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 8 | 6
hours | 8.66 (2.66) | 7.5 (2.49)

6. Primary Outcome: Total Sleep as Assessed by the Misfit Shine Device
Description: as for outcome 4
Time Frame: day 4
Population: Data were not collected for 4 in the suvorexant arm and 4 in the placebo arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 6 | 6
hours | 6.73 (2.19) | 7.39 (2.23)

7. Primary Outcome: Total Sleep as Assessed by the Misfit Shine Device
Description: as for outcome 4
Time Frame: day 7
Population: Data were not collected for one in the suvorexant arm and 4 in the placebo arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 9 | 6
hours | 6.37 (1.91) | 7.5 (1.35)

8. Primary Outcome: Total Sleep as Assessed by the Misfit Shine Device
Description: as for outcome 4
Time Frame: day 9
Population: Data were not collected for 2 in the suvorexant arm and 4 in the placebo arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 8 | 6
hours | 7.91 (1.38) | 8.01 (1.65)

9. Primary Outcome: Total Sleep as Assessed by the Misfit Shine Device
Description: as for outcome 4
Time Frame: day 11
Population: Data were not collected for 4 in the suvorexant arm and 4 in the placebo arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 6 | 6
hours | 6.93 (1.45) | 7.94 (2.73)

10. Primary Outcome: Total Sleep as Assessed by the Misfit Shine Device
Description: as for outcome 4
Time Frame: day 14
Population: Data were not collected for 3 in the suvorexant arm and 5 in the placebo arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 7 | 5
hours | 6.57 (1.96) | 7.56 (0.95)

11. Primary Outcome: Stress as Assessed by the DASS21 Self-report Questionnaire Stress Subscale
Description: DASS21 is a 21-item self-report questionnaire assessing the severity of clinically agreed upon core depression, anxiety, and stress symptoms. It is well validated in multiple languages and countries, and has been utilized in SUD treatment and withdrawal studies. Total score on the stress subscale is 0 to 42, with higher scores indicating worse outcome.
Time Frame: day 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 4.4 (2.84) | 3.8 (3.77)

12. Primary Outcome: Stress as Assessed by the DASS21 Self-report Questionnaire Stress Subscale
Description: as for outcome 11
Time Frame: day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 3.8 (2.44) | 2.5 (2.84)

13. Primary Outcome: Stress as Assessed by the DASS21 Self-report Questionnaire Stress Subscale
Description: as for outcome 11
Time Frame: day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 2.7 (2.31) | 3.1 (4.28)

14. Primary Outcome: Stress as Assessed by the DASS21 Self-report Questionnaire Stress Subscale
Description: as for outcome 11
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.7 (1.7) | 2.7 (3.3)

15. Primary Outcome: Stress as Assessed by the DASS21 Self-report Questionnaire Stress Subscale
Description: as for outcome 11
Time Frame: day 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.9 (2.18) | 2.3 (3.3)

16. Primary Outcome: Stress as Assessed by the DASS21 Self-report Questionnaire Stress Subscale
Description: as for outcome 11
Time Frame: day 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 2 (2.31) | 2.4 (3.24)

17. Primary Outcome: Stress as Assessed by the DASS21 Self-report Questionnaire Stress Subscale
Description: as for outcome 11
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 2.8 (2.66) | 2.3 (4.11)

18. Primary Outcome: Anxiety as Assessed by the DASS21 Self-report Questionnaire Anxiety Subscale.
Description: DASS21 is a 21-item self-report questionnaire assessing the severity of clinically agreed upon core depression, anxiety, and stress symptoms. It is well validated in multiple languages and countries, and has been utilized in SUD treatment and withdrawal studies. Total score on the anxiety subscale is 0 to 42, with higher scores indicating worse outcome.
Time Frame: day 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 2.6 (1.84) | 2.3 (2)

19. Primary Outcome: Anxiety as Assessed by the DASS21 Self-report Questionnaire Anxiety Subscale
Description: as for outcome 18
Time Frame: day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.9 (2.02) | 2.1 (2.28)

20. Primary Outcome: Anxiety as Assessed by the DASS21 Self-report Questionnaire Anxiety Subscale
Description: as for outcome 18
Time Frame: day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.5 (2.12) | 1.4 (1.65)

21. Primary Outcome: Anxiety as Assessed by the DASS21 Self-report Questionnaire Anxiety Subscale
Description: as for outcome 18
Time Frame: day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.5 (2.42) | 1.2 (1.48)

22. Primary Outcome: Anxiety as Assessed by the DASS21 Self-report Questionnaire Anxiety Subscale
Description: as for outcome 18
Time Frame: day 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.4 (2.32) | 0.9 (1.1)

23. Primary Outcome: Anxiety as Assessed by the DASS21 Self-report Questionnaire Anxiety Subscale
Description: as for outcome 18
Time Frame: day 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 1.4 (1.9) | 0.8 (1.03)

24. Primary Outcome: Anxiety as Assessed by the DASS21 Self-report Questionnaire
Description: as for outcome 18
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 2.2 (2.49) | 1.1 (1.6)

25. Secondary Outcome: Cue Reactivity as Assessed by the Cocaine Craving Questionnaire (CCQ) Brief
Description: The Cocaine Craving Questionnaire (CCQ) Brief is a self-report, 14-item measure with five conceptual domains: Desire to Use, Intention to Use, Anticipation of Positive Outcome, Anticipation of Relief from Dysphoria, and Lack of Control over use. The measure is well validated and has been used in multiple studies of CUD. Total score ranges from 1 to 7. A higher score indicates a worse outcome.
Time Frame: day 0, day 7, and day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  day 0 | 3.61 (1.24) | 2.7 (1.26)
  day 7 | 3.01 (1.3) | 2.8 (1.02)
  day 14 | 2.92 (1.47) | 2.48 (0.98)

26. Secondary Outcome: Sleep Quality as by the Pittsburg Sleep Quality Index (PSQI)
Description: The Pittsburg Sleep Quality Index (PSQI) is an 18-item self-report measure of sleep, providing a well-validated and reliable measure of sleep quality, latency, duration, duration efficiency, and disturbance, and an overall summary. The overall summary score will be reported for this measure. The PSQI has been used in several studies of individuals with SUD, including cocaine. Total score ranges from 0-21, with a higher score indicating worse outcome.
Time Frame: day 0, day 2, day 4, day 7, day 9, day 11, and day 14
Population: Data were not collected for days 2, 4, 9, and 11. For days 0, 7, and 14, where number analyzed is less than 10, data were not collected for the number that are not reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  day 0 | 7.5 (2.46) | 7 (2.36)
  day 2: number analyzed (Participants) | 0 | 0
  day 4: number analyzed (Participants) | 0 | 0
  day 7: number analyzed (Participants) | 8 | 10
  day 7 | 9.38 (4.24) | 6.6 (2.91)
  day 9: number analyzed (Participants) | 0 | 0
  day 11: number analyzed (Participants) | 0 | 0
  day 14: number analyzed (Participants) | 10 | 9
  day 14 | 8.2 (3.19) | 4.89 (1.76)

27. Secondary Outcome: Stress/Anxiety as Assessed by Blood Pressure During the Cold Pressor Test (CPT) - Systolic Blood Pressure
Description: Cold Pressor Test (CPT) reliably increases activity of the sympathetic nervous system and the HPA axis, and produces reliable increases in heart rate and cortisol. Subjects are requested to submerge the dominant arm up to the wrist or elbow in ice-cold water (0° to 4° C) for as long as possible with a maximum of 90 seconds. The procedure activates afferent nerves and elicits a CNS stress response. This procedure produces no lasting biological or psychological distress beyond the acute challenge period, and physiological effects return to baseline within 90 min. In fact, the CPT is used to study pain in children, and is considered a noninvasive, exempt educational experimental activity by the IRB of the University of Texas-Austin. It has been used extensively in cardiology, endocrinology, psychiatry, and psychology since 1940 as a challenge to the peripheral and central stress axis
Time Frame: day 0, day 7, and day 14
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
millimeters of mercury (mmHg)
  day 0, immediately before CPT | 125 (12.9) | 120 (17.4)
  day 7, immediately before CPT | 126 (10.3) | 125 (16.1)
  day 14, immediately before CPT | 128 (17.7) | 121 (16.6)
  day 0, immediately after CPT | 123 (12.3) | 113 (13.5)
  day 7, immediately after CPT | 122 (12.2) | 132 (19.3)
  day 14, immediately after CPT | 120 (15.8) | 120 (20)

28. Secondary Outcome: Stress/Anxiety as Assessed by Blood Pressure During the Cold Pressor Test (CPT) - Diastolic Blood Pressure
Description: as for outcome 27
Time Frame: day 0, day 7, and day 14
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
millimeters of mercury (mmHg)
  day 0, immediately before CPT | 84.6 (9.43) | 80.7 (17.4)
  day 7, immediately before CPT | 84.8 (10.5) | 83.6 (12)
  day 14, immediately before CPT | 85.4 (12.9) | 81.1 (10)
  day 0, immediately after CPT | 82 (8.51) | 72.3 (9.1)
  day 7, immediately after CPT | 82.6 (9.34) | 87.2 (13.1)
  day 14, immediately after CPT | 76.3 (19.3) | 80.2 (12.4)

29. Secondary Outcome: Stress/Anxiety as Assessed by Cortisol Level During the Cold Pressor Test (CPT)
Description: as for outcome 27
Time Frame: day 0, day 7, and day 14
Population: Where number analyzed is less than 10, data were not collected for the number that are not reported.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
pg/mL
  day 0, immediately before CPT: number analyzed (Participants) | 10 | 9
  day 0, immediately before CPT | 553 (291) | 1269 (2070)
  day 7, immediately before CPT: number analyzed (Participants) | 9 | 9
  day 7, immediately before CPT | 1108 (690) | 957 (1211)
  day 14, immediately before CPT: number analyzed (Participants) | 7 | 10
  day 14, immediately before CPT | 532 (522) | 629 (391)
  day 0, immediately after CPT: number analyzed (Participants) | 10 | 9
  day 0, immediately after CPT | 582 (448) | 894 (377)
  day 7, immediately after CPT: number analyzed (Participants) | 9 | 9
  day 7, immediately after CPT | 873 (904) | 1280 (2063)
  day 14, immediately after CPT: number analyzed (Participants) | 7 | 10
  day 14, immediately after CPT | 589 (286) | 1120 (770)

30. Secondary Outcome: Stress as Assessed by a Visual Analog Scale (VAS) for Stress
Description: Score provided is the total score (0 to 300) across three items that are each on a 0-100 scale. A higher score indicates greater stress.
Time Frame: day 0, day 2, day 4, day 7, day 9, day 11, and day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  day 0 | 192 (44.1) | 138 (63)
  day 2 | 168 (54.8) | 127 (52.6)
  day 4 | 151 (80.5) | 124 (53.2)
  day 7 | 128 (50.1) | 134 (75.4)
  day 9 | 145 (45.9) | 118 (66.3)
  day 11 | 145 (54.9) | 142 (66.2)
  day 14 | 142 (79.4) | 119 (76.4)

31. Secondary Outcome: Percent Medication Compliance as Assessed by the Medical Event Monitoring System (MEMS, Aprex Corporation) Bottles
Time Frame: day 2, day 4, day 7, day 9, day 11, and day 14
Measure: Mean (Standard Deviation); unit: percent medication compliance
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
percent medication compliance
  day 2 | 91.9 (0.302) | 100 (0)
  day 4 | 81.8 (0.405) | 100 (0)
  day 7 | 81.8 (0.405) | 100 (0)
  day 9 | 81.8 (0.405) | 100 (0)
  day 11 | 100 (0) | 75 (0.463)
  day 14 | 81.8 (0.405) | 87.5 (0.354)

32. Secondary Outcome: Percent Medication Compliance as Assessed by Pill Counts
Time Frame: day 2, day 4, day 7, day 9, day 11, and day 14
Measure: Mean (Standard Deviation); unit: percent medication compliance
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
percent medication compliance
  day 2 | 95.5 (0.151) | 100 (0)
  day 4 | 95 (0.158) | 100 (0)
  day 7 | 100 (0) | 100 (0)
  day 9 | 100 (0) | 88.9 (0.333)
  day 11 | 90 (0.316) | 100 (0)
  day 14 | 100 (0) | 100 (0)

33. Secondary Outcome: Percent Medication Compliance as Assessed by Analysis of Riboflavin Markers in Urine Samples
Time Frame: day 2, day 4, day 7, day 9, day 11, and day 14
Measure: Mean (Standard Deviation); unit: percent medication compliance
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
percent medication compliance
  day 2 | 100 (0) | 100 (0)
  day 4 | 100 (0) | 89 (0.333)
  day 7 | 100 (0) | 100 (0)
  day 9 | 100 (0) | 100 (0)
  day 11 | 90 (0.316) | 100 (0)
  day 14 | 100 (0) | 100 (0)

34. Secondary Outcome: Percent Medication Compliance as Assessed by Text Reminders and Replies
Description: Text-based reminders to take the medication will be enabled via using a HIPAA secure texting service (Talksoft ©), used broadly in medical settings. Participants will be prompted each night at 10 PM to take their medication, and instructed to text back "yes" when they have taken their medication.
Time Frame: day 2, day 4, day 7, day 9, day 11, and day 14
Measure: Mean (Standard Deviation); unit: percent medication compliance
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
percent medication compliance
  day 2 | 55.6 (0.527) | 100 (0)
  day 4 | 55.6 (0.527) | 87.5 (0.354)
  day 7 | 70 (0.483) | 100 (0)
  day 9 | 70 (0.483) | 100 (0)
  day 11 | 90 (0.316) | 75 (0.463)
  day 14 | 87.5 (0.354) | 75 (0.463)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02785406/Prot_SAP_000.pdf